CLINICAL TRIAL: NCT06833619
Title: Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Elbadry Elrabie, Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-12---6MD
Record Dates: First submitted 2024-12-18; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique (Other)
  Interventions: Device: Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique

INTERVENTIONS:
Device: Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique — Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique

SUMMARY:
Endoscopic ultrasound-guided liver biopsy (EUS-LB) can overcome many shortcomings of percutaneous liver biopsy and TJLB. Targeted and non-targeted liver biopsies can be done through this biopsy. It can be done in patients with international normalized ratio (INR) up to 2. It has less tissue fragmentation compared with TJLB.

Needle entering the liver can be viewed in real-time (intrahepatic vessels and bile duct can be spared from injury) (Sharma et al., 2023). Both lobes of the liver can be accessed. It provides minimal patient discomfort. EUS-LB can access liver lesions that may not be safely accessible by routine US or computed tomography (tenBerge et al., 2002). It provides better results in obese individuals compared with percutaneous liver biopsy. It is safe in pregnant females requiring liver biopsy (Khare et al., 2024). Despite these advantages, EUS-LB is largely limited to tertiary care centers and its use is not yet widespread. This may be because, since its inception, numerous variations in needle shape, needle size, and, most notably, sampling techniques have been adopted.

However, no consensus protocol for acquisition has been recognized, leading to poor procedural standardization and wide ranges of reported outcomes in sample quality and diagnostic yield. As such, there is a substantial need for a uniform technique that will safely maximize diagnostic performance with minimal needle passes (Khare et al., 2024).

ELIGIBILITY:
Inclusion Criteria:

* The participants of the study were adults in need of liver biopsy for the evaluation of Altered liver function test

Exclusion Criteria:

* Using anti-platelets or anticoagulants within the last 5days
* Inability to provide informed consent
* Moderate-to-gross ascites
* Child C cirrhosis
* INR more than 2.01
* Platelet count less than 50,000/µL3

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Endoscopic Ultrasound Guided Liver Biopsy Using Dynamic Wet Technique | -Study period: Duration of the study will be 12 months after acceptance of The Ethical Committee Of The Medical Research. All patients will sign an informed written consent before starting the data collection with respect to patient's confidentiality.
  Measurement the efficacy of liver biopsy specimens by European Association for the Study of Liver Disease (EASL) criteria .
  - Total Specimen Length (TSL) of more than or equal to 15 mile-meters.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Elbadry Eirabie, master, Study Director — Sohag
Locations (1):
- Sohag University, Sohag, Egypt